CLINICAL TRIAL: NCT03811470
Title: China Diabetes Registry - a Prospective Cohort Study of Patients With Diabetes in National Metabolic Management Centers in China
Brief Title: China Diabetes Registry by Metabolic Management Center
Acronym: CDR-MMC
Status: Recruiting | Type: Observational
Sponsor: Guang Ning (Other)
Responsible Party: Sponsor-Investigator, Guang Ning, Vice-president of Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Chairman of the Chinese National Clinical Research Center for Endocrine and Metabolic Diseases, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: CCEMD-2018-1201
Record Dates: First submitted 2018-12-20; First posted 2019-01-22 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes Mellitus; Type1 Diabetes Mellitus; Monogenetic Diabetes; Pancreatogenic Diabetes; Drug-Induced Diabetes Mellitus; Other Forms of Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — DNA, Serum, plasma and full blood samples are retained
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with diabetes mellitus including: type 1 or type 2 diabetes mellitus, monogenetic diabetes, pancreatogenic diabetes, drug-induced diabetes, other forms
  Interventions: Other: Standard diabetes management model in each MMC center

INTERVENTIONS:
Other: Standard diabetes management model in each MMC center — Standard diabetes management model in each MMC center

SUMMARY:
Epidemiologic studies have revealed a tremendous increase in the prevalence of diabetes and related mortality worldwide. In order to meet all the challenges in the treatment of metabolic diseases in China, the National Metabolic Management Center (MMC) was founded in 2016. The objective of the MMC is to launch a new metabolic disease management model based on the Internet health information platform. It allows the application and evaluation of diabetes treatment strategies at these centers. The proprietary electronic medical database in the MMC will help the dynamic big-data analysis in diabetes epidemiology, prevention, diagnosis, and treatment. It will also provide prospective data support including economic evaluation in management of chronic diseases for the Healthy China 2030 strategy.

Objective

1. The purpose of the present study is to establish a multi-center nationwide prospective database of diabetes patients in MMCs, including clinical data, biological samples library so as to explore the epidemiology, genetics, new biomarkers, risk factors, and prognostic methods related to diabetes and its complications, as well as other metabolic diseases.
2. To collect cross-sectional data from patients seen and treated at each MMC centers so as to evaluate: the current status of care of patients with diabetes and its related complications, as well as other risk factors treatment strategies at these centers. Patients'costs and quality of life (QoL) will also be evaluated.
3. To collect the prospective data of patients treated at each MMC centers in order to evaluate the strategies for the achievement of treatment goals, changes in management, control of risk factors, incidence and progression of all-diabetes related clinical endpoints (including mortality), behavioral changes, psychological well being as well as costs and QoL.

DETAILED DESCRIPTION:
Epidemiologic studies have revealed a tremendous increase in the prevalence of diabetes and related mortality worldwide. The general population-based survey in China in 2010, using the American Diabetes Association (ADA) 2010 criteria, revealed that the prevalence of diabetes and prediabetes in adults was 11.6% and 50.1%, respectively, indicating that China has the highest diabetes prevalence in Asia and largest absolute disease burden of diabetes in the world. Lifestyle changes, aging, and obesity have become the main reasons for this increase in the prevalence of diabetes.

In order to meet all the challenges in the treatment of metabolic diseases in China, the National Metabolic Management Center (MMC) was founded in 2016. With advanced medical equipment and Internet of Things (IoT) technology, the MMC is committed to creating an online and offline integrated solution for diabetes, and for the entire spectrum of metabolic disease, to achieve a more convenient and precise model of care for patients. The MMC is focused on establishing highly efficient diagnosis and treatment, as well as comprehensive disease management both in and out of hospital. All MMCs in China have the same structure in terms of facilities, layout, and databases, as well as the same routine daily operations, aiming to establish a platform with standardized diagnosis and treatment of metabolic diseases and their long-term follow-up. This platform of treatment is called the'One Center, One Stop, and One Standard Model'.

The objective of the MMC is to launch a new metabolic disease management model based on the Internet health information platform. It allows the application and evaluation of diabetes treatment strategies at these centers. The proprietary electronic medical database in the MMC will help the dynamic big-data analysis in diabetes epidemiology, prevention, diagnosis, and treatment. It will also provide prospective data support including economic evaluation in management of chronic diseases for the Healthy China 2030 strategy.

Objective：

1. The purpose of the present study is to establish a multi-center nationwide prospective database of diabetes patients in MMCs, including clinical data, biological samples library so as to explore the epidemiology, genetics, new biomarkers, risk factors, and prognostic methods related to diabetes and its complications, as well as other metabolic diseases.
2. To collect cross-sectional data from patients seen and treated at each MMC centers so as to evaluate: the current status of care of patients with diabetes and its related complications, as well as other risk factors treatment strategies at these centers. Patients'costs and quality of life (QoL) will also be evaluated.
3. To collect the prospective data of patients treated at each MMC centers in order to evaluate the strategies for the achievement of treatment goals, changes in management, control of risk factors, incidence and progression of all-diabetes related clinical endpoints (including mortality), behavioral changes, psychological well being as well as costs and QoL.

Methods： After obtaining informed consent, patients will be invited and initiated with a comprehensive baseline evaluation at each MMC centers. Then patients will be followed by clinical/laboratory visits at MMC every 3-6 month later on according to individualized patient's treatment plans. A repeated comprehensive clinical and laboratory assessment for glycemic and risk factors control, safety, as well as diabetes-specific complications will be scheduled once a year.

ELIGIBILITY:
Main Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of diabetes mellitus based on self-reported history of diagnosed diabetes by clinicians or in line with the current domestic diagnostic criteria for diabetes
* Gender: males and females
* Provide written informed consent
* Satisfactory compliance

Main Exclusion Criteria:

* Patients with significantly reduced life expectancy (less than 5 years)
* With Drug abuse
* With AIDS or syphilis or infectious diseases such as viral hepatitis or tuberculosis in active phase at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients who are seen and treated at each MMC centers, and meet the In-/Ex-clusion Criteria will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2037-05-31 (Estimated); Study Completion 2039-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of all diabetes-related clinical endpoints; including: 1. Macrovascular morbidity | through study completion, up to 20 years
Microvascular morbidity | through study completion, up to 20 years
Mortality | through study completion, up to 20 years
Major infections - pulmonary and non-pulmonary requiring hospitalizations | through study completion, up to 20 years
Heart failure | through study completion, up to 20 years
  including hospitalized or treated heart failure, or heart failure death
Neuropathy | through study completion, up to 20 years
  defined as a composite score by the assessment of positive responses among symptoms (by a careful history), sensory signs, or absent or hypoactive reflexes consistent with a distal symmetrical polyneuropathy, and at least one abnormal nerve conduction
All cancers | through study completion, up to 20 years
  The occurrence of any of the following cancers: prostate, breast, lung/bronchus, endometrial, colon, gastric, leukemia, lymphoma, pancreas, kidney/renal pelvis, rectal, and melanoma, etc

SECONDARY OUTCOMES:
HbA1c (%) | through study completion, up to 20 years
Fasting and postprandial glucose (mmol/L) | through study completion, up to 20 years
Blood pressures (mmHg) | through study completion, up to 20 years
lipids (mg/dl) | through study completion, up to 20 years
Body mass index (BMI) | through study completion, up to 20 years
  Body weight (kg) and height (m) will be combined to report BMI in kg/m^2
Visceral fat (cm^2) | through study completion, up to 20 years
Health related quality of life | through study completion, up to 20 years
  Evaluated with HQoL scales such as Short Form 12 Health Survey Questionnaire
Cognitive function | through study completion, up to 20 years
  Incidences of all-cause dementia and mild cognitive impairment, cognitive function assessed by cognitive function scale
Psychological well being | through study completion, up to 20 years
  using physiological parameter, questionnaire
Cost-effectiveness | through study completion, up to 20 years
  The incremental cost per quality adjusted life year (QALY) gained. QALYs will be measured by the EuroQol-5 Dimensions (EQ-5D) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- National Metabolic Management center, Multiple Locations, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang Y, Wang W, Ning G. Metabolic Management Center: An innovation project for the management of metabolic diseases and complications in China. J Diabetes. 2019 Jan;11(1):11-13. doi: 10.1111/1753-0407.12847. Epub 2018 Oct 3. No abstract available. PMID 30284373
- [Derived] Mu L, Li C, Zhao W, Li A, Zhao D, Zhang B. Association between Sleep Duration and Left Ventricular Hypertrophy for Patients with Type 2 Diabetes Mellitus. Int J Endocrinol. 2023 Nov 28;2023:5532778. doi: 10.1155/2023/5532778. eCollection 2023. PMID 38131034
- [Derived] Li L, Mi Y, Xu M, Ruan L, Sun J, Song Q. Influence of Dietary Salt Intake on T2D Treatment. Front Endocrinol (Lausanne). 2022 Jun 15;13:926143. doi: 10.3389/fendo.2022.926143. eCollection 2022. PMID 35784580
- [Derived] Yang X, Lin Y, Xu GD, Chen YS, Zhou Y, Sun J, Li L. Optimal Cut-Off Values of Visceral Fat Area for Predicting Metabolic Syndrome Among Type 2 Diabetes Patients in Ningbo, China. Diabetes Metab Syndr Obes. 2021 Mar 25;14:1375-1383. doi: 10.2147/DMSO.S304164. eCollection 2021. PMID 33790605

DOCUMENTS (1):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03811470/Prot_000.pdf